CLINICAL TRIAL: NCT00438087
Title: Assessment of Corticosteroid Effect in the Prevention of Facial Palsy After Cerebella-pontine Angle Surgery
Brief Title: Corticosteroids in Prevention of Facial Palsy After Cranial Base Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P051072
Record Dates: First submitted 2007-02-09; First posted 2007-02-21 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Facial Palsy
Keywords: Facial palsy; Vestibular schwannoma; Anti-inflammatory drugs; Post surgery of vestibular schwannoma; or of cranial base tumors
MeSH Terms: conditions — Facial Paralysis; Neuroma, Acoustic | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): placebo versus methylprednisolone
  Interventions: Drug: methylprednisolone
- 1 (Experimental): placebo versus methylprednisolone
  Interventions: Drug: methylprednisolone

INTERVENTIONS:
Drug: methylprednisolone — methylprednisolone administrated intra and post operatively
  Other Names: methylprednisolone administrated intra and post operatively

SUMMARY:
Facial palsy after surgical removal of cranial base tumors adherent to the nerve can partly be explained by inflammation.

DETAILED DESCRIPTION:
Facial palsy after surgical removal of cranial base tumors adherent to the nerve can partly be explained by inflammation.

The purpose of this study was to assess the efficiency of corticosteroids to prevent facial palsy after such surgery and to identify the patients that will have the highest benefit from an anti-inflammatory treatment.

This study will include patients undergoing surgery for a benign tumor of the cranial base (vestibular schwannoma). The efficiency of high dosage corticosteroids administered intravenously during and after surgery will be evaluated on the facial nerve function in comparison to a placebo. Pre operative and intra operative data will be collected and analysed in order to investigate possible predictive factors of response to the treatment.

Introduction: After the surgical removal of a cerebella-pontine angle tumor (mainly vestibular schwannoma), and despite the anatomical integrity of the facial nerve, an immediate or delayed facial palsy may occur. This palsy may be explained by ischemia, edema, inflammation, or a neurotmesis (ruptured axons in an intact nerve sheet). This phenomenon is highly dependent on the size of the tumor. In our preliminary studies, we observed an immediate facial palsy in 16% and a palsy occurring at postoperative day 8 in 23% of the patients operated on for a vestibular schwannoma. Corticosteroids may decrease the inflammation and the edema around the nerve and reduce the incidence of the postoperative facial palsy. Their efficiency has already been demonstrated in idiopathic facial palsy. In a previously published study , a single dose of dexamethasone during surgery did not influence the facial function outcome. But the short period of the treatment do not allow definitive conclusions.

Objectives: The aim of this study is to analyze the effect of a corticosteroid (methyl prednisolone) administered intra- and postoperatively on the incidence of facial palsy after surgery of cerebella-pontine angle tumors and to determine intra operative prognostic factors for the facial function outcome.

Material and Methods: A multi center, prospective, randomized, versus placebo, and double-blind study will be undertaken. Four-hundred patients undergoing surgery for a cerebellopontine angle tumor will be included during 23 months. Three university departments of otolaryngology (Hospital BEAUJON, CHU de Bordeaux, CHU de Tours) will participate. The pre operative assessment includes a clinical examination with the assessment of the facial function (in 6 grades according to House and BRACKMANN), an audiometry and a vestibular testing, and a cranial MRI with the classification of tumors in 4 stages according to their size. Patients will be randomized after information and with their consent. During surgery, the degree of nerve stretch (4 stages), the tumor adhesion to the nerve (4 stages) and the stimulation thresholds of the facial nerve with an electromyographic monitoring device (NIM Response 2, XOMED MEDTRONICS, Jacksonville, FL) will be recorded. All cases of facial nerve interruption during surgery will be excluded. In the treated group, one IV injection of methyl prednisolone at 1 mg/kg/day will be administered intra operatively and on postoperative days 1 and 2. The treatment will be continued on days 3 to 7 with the same dosage orally. Subsequently, 0.5 mg/kg/day at days 8 and 8, and 0.25 mg/kg/day at days 10 and 11. The facial function will be assessed on postoperative days 1, 8 and 30 clinically.

Expected results: Considering the effect of corticosteroids in the idiopathic facial palsy and the effect of these agents on edema and inflammation, we expect and decrease in the incidence of immediate and delayed postoperative facial palsies. The intra operative stimulation thresholds may indicate a subgroup of patients for which the efficiency of the corticosteroids is higher than in the whole series.

Conclusion : The facial palsy after surgery of cerebellopontine angle tumors is the most frequent and the most significant morbidity. Corticosteroids may decrease the incidence of this complication.

ELIGIBILITY:
Inclusion Criteria:

* adults patients
* surgery of base crane tumors
* accept to participate
* having health insurance

Exclusion Criteria:

* pregnant woman
* children
* known allergy to steroids
* preoperative facial palsy of grade >2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2007-03; Primary Completion 2010-03 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the facial function at 8 days postoperative | at 8 days postoperative

SECONDARY OUTCOMES:
Assessment of the facial function at 1 day postoperative | at 1 day postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Alexis BOZORG GRAYELI, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Assistance Publique Hopitaux de Paris, Clichy, France